CLINICAL TRIAL: NCT07183917
Title: Forest Therapy and Mindfulness for Stress Reduction and Well-being in Highly Sensitive Persons: A Randomized Controlled Pilot Trial
Brief Title: "Forest Therapy and Mindfulness for Stress Reduction and Well-being in Highly Sensitive Persons (Pilot RCT)"
Acronym: HSP-FOREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IFM International Forest Medicine (Other)
Responsible Party: Principal Investigator, Ana I. Sánchez Hdz., "Dr. Ana I. Sánchez Hdz., Sponsor-Investigator, IFM International Forest Medicine, responsible for study design, implementation, and compliance with ethical and clinical research standards.", IFM International Forest Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSP-FOREST-2025-RCT
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

Keywords: Forest Bathing; Shinrin-Yoku; Forest Therapy; Highly Sensitive Person (HSP); Integrative Medicine; Preventive Health; Psychological Well-Being; Nature Therapy; Mindfulness; Stress Reduction; Mental healht; Forest meicine
MeSH Terms: conditions — Psychological Well-Being | interventions — Forest Therapy; Mindfulness

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group randomized controlled design with 1:1 allocation. Participants are assigned to (a) Forest Therapy + Mindfulness or (b) Indoor Wellness Activities (active control). No crossover is planned. The intervention spans 8 weeks with weekly 2-hour group sessions. Randomization uses a computer-generated sequence with concealed allocation (sealed, opaque envelopes), block sizes of 4-6, and stratification by sex and baseline PSS-10 (median split). Open-label for participants and providers; outcomes assessors/statisticians remain blinded to group codes during analysis.
Masking Description: Due to the nature of the intervention (forest therapy and mindfulness), blinding is not feasible. This study uses an open-label design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Forest Therapy + Mindfulness (Experimental): Weekly 2-hour guided sessions for 8 weeks in natural forest environments, including mindful walking, sensory awareness, breathing exercises, and guided relaxation.
  Interventions: Behavioral: Forest Therapy and Mindfulness
- Active Comparator: Indoor Wellness Activities (Active Comparator): Weekly 2-hour indoor sessions for 8 weeks in a classroom or community center setting, including health education talks, guided relaxation or music therapy, and eco-culinary tasting.
  Interventions: Behavioral: Indoor Wellness Control

INTERVENTIONS:
Behavioral: Forest Therapy and Mindfulness — Weekly 2-hour guided sessions for 8 consecutive weeks in natural forest environments. Each session includes mindful walking, multisensory awareness (sight, sound, smell, touch), breathing exercises, and guided relaxation practices. Facilitated by certified Forest Therapy and Mindfulness instructors. The intervention is non-invasive, focused on stress reduction, emotional regulation, and improved subjective well-being through mindful immersion in nature.
  Arms: Experimental: Forest Therapy + Mindfulness
Behavioral: Indoor Wellness Control — Weekly 2-hour structured sessions for 8 consecutive weeks conducted indoors (classroom or wellness center). Activities include health education talks on stress and wellness, guided music-based relaxation, and eco-friendly culinary tasting experiences. Designed to provide an active comparator condition controlling for attention, group interaction, and wellness-related content without exposure to forest environments or formal mindfulness practices.
  Arms: Active Comparator: Indoor Wellness Activities

SUMMARY:
This study aims to evaluate the effects of Shinrin-Yoku (Forest Bathing) and Forest Medicine interventions on psychological well-being, stress reduction, and overall health outcomes in adults. Shinrin-Yoku, originated in Japan, is a nature-based practice that involves mindful immersion in forest environments. The intervention combines exposure to natural ecosystems with evidence-based techniques such as mindfulness and guided relaxation.

Participants will be guided through structured sessions in natural forest settings to assess changes in stress biomarkers, emotional regulation, sleep quality, and quality of life. The study is designed as a non-pharmacological, non-invasive intervention, focusing on promoting mental health and preventive medicine.

The findings are expected to provide evidence on the benefits of Forest Medicine as a complementary health approach and contribute to the development of international standards for nature-based therapies.

DETAILED DESCRIPTION:
The present study investigates the therapeutic potential of Shinrin-Yoku (Forest Bathing) and Forest Medicine interventions as structured nature-based health practices. Originating in Japan during the 1980s, Shinrin-Yoku has gained recognition worldwide for its reported psychological and physiological benefits. This research seeks to contribute to the scientific evidence supporting these interventions as complementary approaches in preventive and integrative medicine.

Participants will attend guided sessions in natural forest environments. Each session will include periods of mindful walking, sensory awareness exercises, and guided relaxation. No pharmacological or invasive procedures are involved. Outcome measures include validated psychological scales (e.g., stress, anxiety, depression, quality of life), as well as physiological indicators such as heart rate variability and sleep quality.

The study design follows an interventional model focusing on mental health and wellness promotion. Data collection will be conducted before, during, and after the intervention period to assess both immediate and sustained effects.

This project is intended to support the integration of Forest Medicine into broader health strategies, aligning with international research efforts in preventive care, psychosomatic health, and nature-based therapeutic modalities. The study also aims to establish standards for training and best practices in forest-based health interventions across Europe and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Self-identified as Highly Sensitive Person (HSP) with a score ≥70 on the Highly Sensitive Person Scale (HSP-SC).
* Able to attend weekly sessions for 8 consecutive weeks.
* Willing to provide written informed consent.

Exclusion Criteria:

* Current diagnosis of severe psychiatric disorder (e.g., schizophrenia, bipolar disorder not stabilized).
* Current substance abuse or dependence.
* Severe cardiovascular, respiratory, or mobility limitations preventing safe participation in outdoor walking or relaxation exercises.
* Participation in another clinical intervention study during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress (PSS-10) | Baseline and 8 weeks (end of intervention)
  Mean change in Perceived Stress Scale (10-item version, validated questionnaire) scores from baseline to 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: ANA I SÁNCHEZ HDZ, Principal Investigator, Study Chair — ASEUSY - European Association Shinrin Yoku and Forest Medicine -Ana I Sánchez Hdz
Locations (1):
- Sessions conducted in natural forest settings within the Serranía de Ronda, specifically the Valle del Genal area., Ronda, Andalusia, Spain